CLINICAL TRIAL: NCT06794450
Title: Comparison of Recovery Times Between 1 mg/kg Sugammadex and 60 mcg/kg Neostigmine for Moderate Neuromuscular Blockade Induced by Rocuronium in Patients Undergoing Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: Recovery Times of Half Dose Sugammadex and Neostigmine for Rocuronium-induced Neuromuscular Blockade
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AN-202412.01
Record Dates: First submitted 2025-01-13; First posted 2025-01-27 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Neuromuscular Blocking Agents; Reversal of Neuromuscular Blockade; Recovery Time
Keywords: Sugammadex; Neostigmine; recovery time from neuromuscular blockade
MeSH Terms: interventions — Sugammadex; Neostigmine; Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugammadex (Experimental): The subjects in this study were patients underwent laparoscopic cholecystectomy surgery with general anesthesia and muscle relaxant Rocuronium.
  At the end of the surgery, thirty patients will be administered Sugammadex 1 mg/kg as a reversal agent. All patient will receive same anesthetic drug. Patients will be monitored with acceleromyography monitoring tools. Extubation was performed when the Train of Four monitor reached a Train of Four Ratio ≥ 90%.
  Interventions: Drug: Sugammadex 1 mg/kg
- Neostigmine (Active Comparator): The subjects in this study were patients underwent laparoscopic cholecystectomy surgery with general anesthesia and muscle relaxant rocuronium.
  At the end of the surgery, thirty patients will be administered Neostigmine 60 mcg/kg along with 0.4 mg of atropine sulfate per 1 mg of neostigmine as a reversal agent. All patient will receive same anesthetic drug. Patients will be monitored with acceleromyography monitoring tools. Extubation was performed when the Train of Four monitor reached a Train of Four Ratio ≥ 90%.
  Interventions: Drug: Neostigmine + Atropine

INTERVENTIONS:
Drug: Sugammadex 1 mg/kg — Patient in experimental arms will receive i.v. sugammadex 1 mg/kg at the end of operating procedure from the point at which a Train-of-Four Count (TOFC) of 2 is observed
  Arms: Sugammadex
Drug: Neostigmine + Atropine — Patient in active comparators arms will receive i.v. neostigmine 60 mcg/kg along with 0.4 mg of atropine sulfate per 1 mg of neostigmine at the end of operating procedure from the point at which a Train-of-Four Count (TOFC) of 2 is observed
  Arms: Neostigmine

SUMMARY:
In operating procedure with general anesthesia muscle relaxant is usually used to increase success rate of the operation and to give better outcome. The use of reversal drugs aims to reduce the risk of post-operative complications due to muscle relaxants. Neostigmine is commonly used as a reversal drug, but its indirect mechanism of action results in a long and unpredictable recovery time. Sugammadex directly bind and inactivate rocuronium, in which resulting in a faster and predictable recovery time. However, the high price limits the use of sugammadex.

This study aims to compare the effect of half dose sugammadex and neostigmine against the moderate neuromuscular blockade of rocuronium.

The main questions it aims to answer are:

Does half dose sugammadex gives faster recovery time? Researchers will compare sugammadex to neostigmine to see if sugammadex gives faster recovery time.

Participants will:

Be given sugammadex or neostigmine as a reversal drug after the operation done

DETAILED DESCRIPTION:
Neuromuscular blocking agents are frequently utilized to facilitate tracheal intubation, minimize the risk of vocal cord injury, suppress patient movement, and ensure optimal ventilation. The administration of these agents, along with meticulous monitoring of neuromuscular blockade depth, plays a critical role in optimizing the success rates and minimizing complications associated with various surgical procedures, including laparotomy and laparoscopic abdominal surgeries.

At the conclusion of surgery, when muscle relaxation is no longer required, neuromuscular blockade should be reversed promptly, safely, and reliably using appropriate reversal agents to minimize the risk of postoperative complications associated with residual neuromuscular blockade. A study reported that 64% of patients undergoing general anesthesia exhibited a neuromuscular recovery of less than 90% and experienced symptoms of re-curarization in the recovery room.

Various reversal agents are available to counteract the effects of neuromuscular blockade, utilizing either direct or indirect mechanisms of action. Cholinesterase inhibitors, such as neostigmine, are among the most commonly used agents. They act indirectly by inhibiting acetylcholinesterase, thereby preventing the breakdown of acetylcholine at the neuromuscular junction. However, this mechanism is reliant on the individual's acetylcholine production rate, which can limit neostigmine's effectiveness, contributing to its unpredictability, and increase the risk of re-curarization. In contrast, sugammadex is a specialized reversal agent designed specifically to counteract neuromuscular blockade induced by rocuronium. Unlike neostigmine, sugammadex employs a direct mechanism by encapsulating rocuronium molecules and forming an inactive complex. This approach enables a faster onset of action and provides a more consistent and predictable recovery profile.

The utilization of sugammadex in Indonesia remains relatively limited, despite the frequent use of rocuronium as a muscle relaxant. This limited use is largely attributed to the significantly higher cost of sugammadex compared to neostigmine. Nonetheless, research has demonstrated that even at doses lower than the recommended levels, sugammadex achieves faster recovery times compared to neostigmine in reversing neuromuscular blockade induced by rocuronium. This trial looks forward to answering the recovery time of half-dose recommended sugammadex compared with neostigmine with usual dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent laparoscopic cholecystectomy under general anesthesia
* Using muscle relaxant rocuronium
* Aged 18-59 years
* American Society of Anesthesiologists (ASA) physical status classification of 1 or 2.

Exclusion Criteria:

* History of drug allergies to the agents used
* Renal dysfunction
* Musculoskeletal disorders
* Central nervous system disorders
* Difficult airways requiring intubation without the use of muscle relaxants.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Recovery time | 1 hour
  This refers to the duration measured from the point at which a Train-of-Four Count (TOFC) of 2 is observed, indicating the administration of the reversal agent, to the achievement of a Train-of-Four Ratio (TOFR) of 90%.
  Train of four is a electrical stimulus pattern that describe the neuromuscular blockade depth. Acceleromyography device used to monitor the neuromuscular blockade depth. Train of Four count (TOFC) 1-3 counted as moderate neuromuscular blockade, train of count (TOFC) 0 counted as deep neuromuscular blockade, train of four count (TOFC) 4 until train of four ratio (TOFR) 89% counted as mild or minimal neuromuscular blockade, and train of four ratio (TOFR) 90% counted as adequate recovery

SECONDARY OUTCOMES:
Spontaneous recovery time of rocuronium | 3 hours
  This refers to the duration measured from the administration of rocuronium to the achievement of a Train-of-Four Count (TOFC) of 1 and 2
  After administration of rocuronium, subject will undergo deep neuromuscular blockade with train of four count 0. Rocuronium will undergo spontaneous degradation over a certain period, but it depends on the body's response to diffusion, redistribution, metabolism, excretion, and release from the muscle relaxant receptors. The duration from the administration of rocuronium, which causes deep neuromuscular blockade with a TOFC depth of 0, to the achievement of moderate neuromuscular blockade with TOFC depths of 1 and 2 will be measured.
Bradycardia | 1 hour
  Assess the frequency of bradicardia after the reversal agent administered
Hypotension | 1 hour
  Assess the frequency of hypotension (mean arterial pressure under 65) after the administration of reversal agent

CONTACTS AND LOCATIONS:
Overall Officials: Tini T Maskoen, M.D., Study Chair — Faculty of Medicine Universitas Padjadjaran
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia